CLINICAL TRIAL: NCT04090398
Title: Phase II Trial of Radium-223 Dichloride in Combination With Paclitaxel in Patients With Bone Metastatic Breast Cancer
Brief Title: Testing the Addition of Radium Therapy (Radium-223 Dichloride) to the Usual Chemotherapy Treatment (Paclitaxel) for Advanced Breast Cancer That Has Spread to the Bones
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-06088; NCI-2019-06088 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 052001; 10302 (Other: City of Hope Comprehensive Cancer Center LAO); 10302 (Other: CTEP); UM1CA186644 (NIH); UM1CA186716 (NIH)
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic HER2-Negative Breast Carcinoma; Metastatic Malignant Neoplasm in the Bone
MeSH Terms: interventions — Specimen Handling; Magnetic Resonance Spectroscopy; Paclitaxel; Taxes; radium Ra 223 dichloride; X-Rays; Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (paclitaxel, radium Ra 223 dichloride) (Experimental): Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and radium Ra 223 dichloride IV over 1 minute on day 1 of each cycle. Treatment with radium Ra 223 dichloride repeats every 28 days for 6 cycles and treatment with paclitaxel repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan, bone scan and/or MRI, as well as collection of blood samples throughout trial. Patients may optionally undergo SPECT on trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Other: Electronic Health Record Review; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Radiation: Radium Ra 223 Dichloride; Procedure: Single Photon Emission Computed Tomography
- Arm II (paclitaxel) (Active Comparator): Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan, bone scan, and/or MRI, as well as collection of blood samples throughout trial. Patients may optionally undergo SPECT on trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Other: Electronic Health Record Review; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Procedure: Single Photon Emission Computed Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Correlative studies
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Other: Electronic Health Record Review — Ancillary studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Radiation: Radium Ra 223 Dichloride — Given IV
  Other Names: Alpharadin; BAY 88-8223; BAY88-8223; Radium 223 Dichloride; RADIUM RA-223 DICHLORIDE; Radium-223 Chloride; Radium-223 Dichloride; Xofigo
  Arms: Arm I (paclitaxel, radium Ra 223 dichloride)
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; Single-Photon Emission Computed; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; ST; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon

SUMMARY:
This phase II trial studies how well radium-223 dichloride and paclitaxel work in treating patients with advanced breast cancer that has spread to the bones. Radium-223 dichloride is a radioactive drug that behaves in a similar way to calcium and collects in cancer that has spread to the bones (bone metastases). The radioactive particles in radium-223 dichloride act on bone metastases, killing the tumor cells and reducing the pain that they can cause. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving radium-223 dichloride and paclitaxel may work better in treating patients with metastatic breast cancer compared to paclitaxel alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the combination of radium-23 dichloride (radium Ra 223 dichloride) and paclitaxel improves progression-free survival (PFS) compared to paclitaxel alone.

SECONDARY OBJECTIVES:

I. To determine the time to the first symptomatic skeletal event (SSE) (defined as 1st use of radiation therapy to relieve skeletal symptoms, new symptomatic pathologic vertebral or non-vertebral bone fractures, spinal cord compression, or tumor-related orthopedic surgical intervention).

II. To measure the objective response rate (ORR). III. To determine the safety of radium-223 dichloride with paclitaxel. IV. To measure overall survival (OS).

EXPLORATORY OBJECTIVES:

I. To perform molecular profiling assays on malignant and normal tissues, including, but not limited to, whole exome sequencing (WES) and messenger ribonucleic acid (RNA) sequencing (RNAseq), in order to:

Ia. Investigate if molecular alterations in deoxyribonucleic acid (DNA) repair genes are associated with response to radium-223 dichloride, and; Ib. Investigate if loss of heterozygosity in triple negative tumors is associated with response to radium-223 dichloride.

II. To contribute genetic analysis data from de-identified biospecimens to Genomic Data Commons (GDC), a well annotated cancer molecular and clinical data repository, for current and future research; specimens will be annotated with key clinical data, including presentation, diagnosis, staging, summary treatment, and if possible, outcome.

III. To correlate change in level of total alkaline phosphatase, bone-specific alkaline phosphatase, and serum osteocalcin to response to radium-223 dichloride therapy.

IV. To examine the radium-223 dichloride bio-distribution and absorbed dose in each bone metastatic lesions as well as elsewhere in the body including critical organs using dosimetry.

V. To bank formalin-fixed, paraffin-embedded (FFPE) tissue, blood, and nucleic acids obtained from patients at the Experimental Therapeutics Clinical Trials Network (ETCTN) Biorepository at Nationwide Children's Hospital.

VI. To explore the symptomatic adverse events (AE) for tolerability of each treatment arm.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive paclitaxel intravenously (IV) over 1 hour on days 1, 8, and 15 and radium Ra 223 dichloride IV over 1 minute on day 1 of each cycle. Treatment with radium Ra 223 dichloride repeats every 28 days for 6 cycles and treatment with paclitaxel repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) scan, bone scan and/or magnetic resonance imaging (MRI), as well as collection of blood samples throughout trial. Patients may optionally undergo single photon emission computed tomography (SPECT) on trial.

ARM II: Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan, bone scan, and/or MRI, as well as collection of blood samples throughout trial. Patients may optionally undergo SPECT on trial.

After completion of study treatment, patients are followed up at 30 days, then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Women or men with metastatic breast cancer with two or more bone metastases identified by technetium Tc-99m (99mTc) bone scintigraphy and/or CT, at least one of these bone lesions must not have been treated with prior radiation therapy
* A diagnosis of breast cancer must have been histologically or cytologically confirmed at any time point
* Patients with non-bone metastases (in addition to bone metastases) are permitted if:

  * Five or less visceral metastasis (=< 4 cm in size) and asymptomatic (not including lymph nodes)
  * Enlarged lymph nodes =< 4 cm
* Patients with HER2 negative disease (HER2 negativity by immunohistochemistry [IHC] or fluorescent in situ hybridization [FISH] ratio according to the American Society of Clinical Oncology-College of American Pathologists guideline criteria) (Hammond et al., 2010; Wolff et al., 2013). Hormone-receptor positive (estrogen receptor [ER]-positive and/or progesterone receptor [PR]-positive) as well as triple-negative (ER-negative, PR-negative and no overexpression of HER2) breast cancer may be enrolled. Hormone receptor status will be determined at the local institution. ER and PR negativity will be defined as < 1% tumor staining by IHC
* Patient must be eligible to receive therapy with paclitaxel for the treatment of their breast cancer. Patients with hormone-receptor positive disease should have progressed on at least one prior line of hormone therapy and a CDK4/6 inhibitor in the metastatic setting to be eligible (except if patient had a contraindication or intolerable toxicity with the use of these agents). Previous radiation and chemotherapy for the treatment of metastatic breast cancer is allowed
* Age >= 18 years

  * Because no dosing or AE data are currently available on the use of radium-223 dichloride in combination with paclitaxel in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (with the exception of < 3 mg/dL for patients with Gilbert's disease)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN (=< 5 ULN for patients with liver metastasis)
* Creatinine =< 1.5 x institutional ULN OR glomerular filtration rate (GFR) >= 40 mL/min/1.73 m^2
* Hemoglobin > 10 g/dL
* Human immunodeficiency virus (HIV)-infected patients on effective antiretroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, HBV viral load must be undetectable on suppressive therapy if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with asymptomatic, treated brain metastases are permitted if there is no evidence of progression for at least 4 weeks after central nervous system (CNS)-directed treatment, as ascertained by clinical examination or brain imaging (magnetic resonance imaging [MRI] or CT scan) during the screening period
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. History of other active malignancy requiring treatment within the last 3 years or bone marrow dysplasia such as myelodysplastic syndrome (MDS) is not allowed
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association functional classification. To be eligible for this study, patients should be class 2B or better
* Concomitant use of bisphosphonates or denosumab is required (except if medical contraindication such as hypocalcemia or concern for osteonecrosis of the jaw). If not already on bone modifying agents, patient must initiate such therapy within one month before start of study treatment
* The effects of radium-223 dichloride on the developing human fetus are unknown. For this reason and because alpha particle-emitting radiopharmaceutical agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 6 months after the last dose. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Pre-menopausal subjects as well as subjects with ovarian radiation or concomitant treatment with an luteinizing hormone-releasing hormone (LH-RH) agonist/antagonist must have a negative pregnancy test and agree to use an adequate method of contraception as recommended by their treating physicians. Subjects of child-bearing potential who are sexually active and their male partners must agree to utilize, during the treatment period and for 6 months after last dose of radium-223 dichloride, 2 reliable and acceptable methods of contraception used simultaneously: a) barrier method such as a) condoms (male or female) with spermicidal agent or b) diaphragm or cervical cap with spermicide, combined with a highly effective non-hormonal birth control method such as an intra-uterine device. Men treated or enrolled on this protocol must also agree to use adequate contraception and not donate sperm prior to the study, for the duration of study participation, and 6 months after completion of radium-223 dichloride
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible
* No prior paclitaxel in metastatic setting within 2 years prior to radium-223 dichloride start. No prior paclitaxel in adjuvant or neoadjuvant setting within 6 months prior to radium-223 dichloride start

Exclusion Criteria:

* Patients with peripheral neuropathy > grade 1
* Patients who have not recovered from AEs due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who have had chemotherapy or immunotherapy with checkpoint inhibitor within 4 weeks prior to treatment. Patient who receives radiation therapy or hormone therapy within 2 weeks prior to treatment are excluded. For patients on trial therapy prior to study enrollment, washout period of 6 times the half-life of previously administered investigational agents prior to starting radium-223 dichloride is required
* Prior therapy with radionuclides (e.g., strontium, samarium, rhenium, radium)
* Patients who are receiving any other investigational agents. Vaccination for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is allowed as well as any therapy as required for the treatment of active coronavirus disease 2019 (COVID-19) infection
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to radium-223 dichloride or other agents used in study
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because radium-223 dichloride is an alpha particle-emitting radiopharmaceutical agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with radium-223 dichloride, breastfeeding should be discontinued if the mother is treated with radium-223 dichloride. These potential risks may also apply to other agents used in this study
* Imminent/established spinal cord compression, pathological fracture in weight bearing bones or bone lesion with soft tissue component unless treated as appropriate with radiation and/or surgery before starting on trial
* Prior hemibody external radiotherapy
* Patients must not have an active infection requiring systemic treatment
* Patients must not use immunosuppressive medication =< 7 days of registration, EXCEPT for the following:

  * Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection)
  * Systemic corticosteroids at physiologic doses =< 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) is allowed
* Patients with Crohn's disease or ulcerative colitis
* Patients with a marked baseline prolongation of QT/corrected QT interval (QTc) interval (e.g., repeated demonstration of a QTc interval > 480 milliseconds [ms]) (CTCAE grade 1) using Fridericia's QT correction formula
* Patients with a history of additional risk factors for Torsades de Pointes (TdP) (e.g. heart failure, hypokalemia, family history of long QT syndrome)
* The use of concomitant medications that prolong the QT/QTc interval
* Life expectancy < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-08-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From randomization to the first documented tumor progression or death due to any cause, whichever occurred first, assessed up to 2 years
  Tumor progression will be determined from radiographic scans performed every 8 weeks (computed tomography and bone scan) using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. The log-rank test will be used to analyze PFS for comparison of treatment effects, i.e., the only covariate that will be used is the treatment arm. Distributions of PFS times will be estimated using the Kaplan-Meier product-limit method.

SECONDARY OUTCOMES:
PFS | From randomization to the first documented tumor progression or death due to any cause, whichever occurred first, assessed up to 2 years
  Treatment comparison in PFS will be conducted in pre-defined subgroups, including hormone receptor status and presence/absence of visceral metastases and two-sided 80% confidence intervals (CIs) will be provided for each subgroup.
Time to first symptomatic skeletal event (SSE) | From randomization to the occurrence of the first SSE, assessed up to 2 years
  Will be defined as the first use of radiation therapy to relieve skeletal symptoms, new symptomatic pathologic vertebral or non-vertebral bone fractures, spinal cord compression, or tumor-related orthopedic surgical intervention. Distributions of time to SSE will be estimated using the method of Kaplan-Meier and compared between treatment arms using the stratified log-rank test.
Objective response rate | From start of treatment until disease progression, assessed up to 2 years
  Will be defined as the proportion of all subjects with confirmed partial response or complete response according to RECIST 1.1.
Overall survival (OS) | From randomization to death due to any cause, assessed up to 2 years
  The log-rank test will be used as the primary analysis for comparison of treatment effects, i.e., the only covariate that will be used is the treatment arm. Distributions of OS times will be estimated using the Kaplan-Meier product-limit method. The median OS times with two-sided 95% CIs will be estimated for each treatment group.
Incidence of adverse events (AEs) | Up to 30 days after end of study treatment
  Will be assessed by grading all treatment-related AEs and events of clinical interest according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Grade 3 or higher diarrhea or constipation are ECI for the proposed trial. Adverse events will be summarized according to grade, overall and by treatment arm, as number and percentage of participants. All adverse events resulting in discontinuation, dose modification, and/or dosing interruption, and/or treatment delay of drug will also be summarized by treatment arm.

OTHER OUTCOMES:
Molecular profiling assays on malignant and normal tissues | At baseline
  Whole exome sequencing and messenger ribonucleic sequencing will be described qualitatively or quantitatively.

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Malhotra, Principal Investigator — City of Hope Comprehensive Cancer Center LAO
Locations (30):
- United States (30):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Virginia Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2024-09-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT04090398/ICF_000.pdf